CLINICAL TRIAL: NCT04651634
Title: A Phase 2, Randomized, Double-Blind, Placebo Controlled Trial to Evaluate the Safety and Efficacy of MIT-001 in Prevention of Oral Mucositis in Patients Receiving CCRT for Locally Advanced HNSCC
Brief Title: MIT-001 for Prevention of CCRT-Induced OM in HNSCC Patients
Acronym: MIT-001
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: MitoImmune Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: MIT001-OM-01
Record Dates: First submitted 2020-11-26; First posted 2020-12-03 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Oral Mucositis
Keywords: MIT-001; Oral Mucositis; OM; NecroX-7; CCRT-associated OM; CCRT-induced OM; Mitochondria-targeted; ROS scavenger
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Stomatitis

STUDY DESIGN:
Intervention Model Description: The three active treatment groups will receive either 20, 40, and 60 mg/day of MIT-001 IV infusion for 30 minutes, two times per week for 5 to 7 continuous weeks until a cumulative radiation dose of between 60 and 72 Gy, with CCRT. Placebo group will receive placebo, manufactured with the same properties and appearance as MIT 001, at same treatment frequency as MIT-001 with CCRT.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study design will minimize bias and provide reference data (i.e., data from placebo treated subjects) which will aid in the interpretation of results. To limit the occurrence of conscious and unconscious bias in the conduct and interpretation of safety and efficacy results, the study is double blind where the subject, the Investigators/site staff, and the Sponsor staff remain unaware of the treatment assignment. The planned safety assessments that will be performed during the study are considered acceptable measures for ensuring the safety of subjects during a clinical study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- 20 mg (Experimental): MIT-001 20 mg
  Interventions: Drug: MIT-001 plus CCRT
- 40 mg (Experimental): MIT-001 40 mg
  Interventions: Drug: MIT-001 plus CCRT
- 60 mg (Experimental): MIT-001 60 mg
  Interventions: Drug: MIT-001 plus CCRT
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: MIT-001 plus CCRT

INTERVENTIONS:
Drug: MIT-001 plus CCRT — MIT-001 IV-infusion plus CCRT

SUMMARY:
The proposed study in patients with previously untreated locally advanced head and neck squamous cell carcinoma (HNSCC) is designed to evaluate the efficacy and safety of three different doses of MIT-001 compared to the placebo in prevention of oral mucositis (OM) in patients with HNSCC who are undergoing concurrent chemoradiotherapy (CCRT).

DETAILED DESCRIPTION:
Oral mucositis associated with cancer therapy carries a significant morbidity. OM is a common complication in patients receiving CCRT used for treating HNSCC. Mucositis lesions can be painful, affect nutrition and quality of life (QoL), and have a significant economic impact. However, a definitive intervention regime has not been established. Therefore, it is essential to develop appropriate treatment.

MitoImmune Therapeutics Inc. (hereafter referred to as Sponsor) has developed MIT-001 which can scavenge abnormal levels of reactive oxygen species (ROS), enabling the cells to retain mitochondrial membrane permeability and mitochondrial function. This eventually inhibits additional ROS production, indicating that MIT-001 can prevent excessive inflammation caused by ROS. In addition, MIT-001 may possibly 1) block inflammatory cytokine production via inhibiting nuclear factor kappa B (NF kB) or inflammasome dependent pathways, 2) inhibit necrosis/necroptosis via blocking high mobility group box 1 (HMGB1) mediated cytokine production, and 3) balance regulation between T helper type 1/17 (Th1/17) and regulatory T cells.

Based on the pathophysiological progression of CCRT-associated OM, initiated by direct injury to basal epithelial cells which experience deoxyribonucleic acid (DNA) damage and increased ROS levels, Sponsor expects the prevention of OM in patients receiving CCRT of locally advanced HNSCC with MIT 001 by effectively scavenging increased ROS induced by CCRT.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed HNSCC (The American joint committee on cancer [AJCC] 8th edition, Stage II, III, IVA, or IVB), involving either the oral cavity or oropharynx, or HPV-positive Stage I oropharyngeal cancer.
* Treatment plan to receive a continuous course of intensity-modulated radiation therapy (IMRT) for definitive treatment of HNSCC delivered as single daily fractions of 1.8 to 2.5 Gy with a cumulative radiation dose between 60 and 72 Gy (EQD2 of 60 to 72 Gy, α/β ratio=10): Planned radiation treatment fields must include at least 30% of oral cavity that are planned to receive a total of 50 Gy or higher.
* CCRT plan to receive standard cisplatin monotherapy: Standard cisplatin monotherapy administered weekly (30 to 40 mg/m2), once per week for 5 to 7 continuous weeks.
* Eastern Cooperative Oncology Group Performance Status (ECOG-PS) 1 or less
* Serum pregnancy test negative for women of childbearing potential (woman of childbearing potential [WOCBP]

Exclusion Criteria:

* Patients who have active mucositis at screening.
* Planned to receive Erbitux™ (Cetuximab) or other targeted or immune therapy during the study.
* Tumor of the lips, sinuses, or salivary glands or unknown primary tumors.
* Metastatic disease (M1) Stage.
* Known history of severe vascular toxicity or allergies or intolerance to cisplatin and similar platinum-containing compounds.
* Any clinically significant and/or active infection, other systemic illness or condition (other than HNSCC) that would preclude them from participating in the study in the opinion of the Investigator.
* Prior resective surgery (4 weeks or less than 4 weeks from receiving surgery to randomization) for primary tumor under treatment for HNSCC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-06-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of severe OM | From first treatment to 2 months of safety follow-up period after CCRT completion
  severe OM (WHO criteria Grade 3 or higher) at a cumulative radiation dose of 60 Gy

SECONDARY OUTCOMES:
Incidence of OM | From first treatment to 2 months of short-term safety follow-up period after CCRT completion
  Incidence of OM of each Grade (WHO criteria)
Time to onset of severe OM | From first treatment to 2 months of short-term safety follow-up period after CCRT completion
  Time to onset of severe OM, defined as Grade 3 or higher (WHO criteria)
Mouth pain and discomfort | From first treatment to 2 months of short-term safety follow-up period after CCRT completion
  Patient-reported mucositis-related mouth pain and discomfort
Analgesic use for OM | From first treatment to 2 months of short-term safety follow-up period after CCRT completion
  Frequency and Cumulative dose (in morphine mg equivalent)

CONTACTS AND LOCATIONS:
Overall Officials: Jinsang Jung, M.Pharm, Study Director — MitoImmune Therapeutics
Locations (16):
- United States (6):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Norris Comprehensive Cancer Center, Los Angeles, California
  - Cancer Center of Kansas, Wichita, Kansas
  - James P. Wilmot Cancer Center, Rochester, New York
  - Wake Forest Baptist Health - Comprehensive Cancer Center, Winston-Salem, North Carolina
  - James Cancer Hospital Solove Research Institute, Columbus, Ohio
- South Korea (10):
  - The Catholic University of Korea Saint Vincent's Hospital, Suwon, Gyeonggi-do
  - Jeonbuk National University Hospital, Jeonju, Jeollabuk-do
  - Keimyung University Dongsan Hospital, Daegu
  - Chungnam National University Hospital, Daejeon
  - National Cancer Center, Goyang-si
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Inha University Hospital, Incheon
  - Seoul National University Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Hanyang University Seoul Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No